CLINICAL TRIAL: NCT00130936
Title: Combined Phase I/II Study of Epirubicin (Pharmorubicin®), Carboplatin (Paraplatin®) and Capecitabine (Xeloda®) (ECC) in the Treatment of Unresectable Locally Advanced or Metastatic Gastric/Gastroesophageal Junction Cancer With Pharmacogenetic Correlates
Brief Title: Study of Epirubicin (Pharmorubicin®), Carboplatin (Paraplatin®) and Capecitabine (Xeloda®) (ECC) in the Treatment of Unresectable Locally Advanced or Metastatic Gastric/Gastroesophageal Junction Cancer With Pharmacogenetic Correlates
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI-05-0046
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2009-09

CONDITIONS: Gastric Cancer; Esophageal Cancer; Tumors
Keywords: phase I; epirubicin; solid tumors
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Neoplasms | interventions — Epirubicin; Carboplatin; Capecitabine

INTERVENTIONS:
Drug: Epirubicin
Drug: Carboplatin
Drug: Capecitabine

SUMMARY:
Although declining in incidence, gastric/gastroesophageal cancer is still a commonly diagnosed malignancy in Canada. Patients who have undergone surgical resection for early disease have a high rate of local recurrence and distant spread. More than 50% of patients present with either locally advanced or metastatic disease. Patients with advanced disease have an extremely poor prognosis, with average survival times ranging from 3 - 9 months. Development of new therapeutic approaches for locally advanced or metastatic gastric/gastroesophageal cancer, is clearly needed.

Despite its proven efficacy, ECF (epirubicin, cisplatin, and infusional 5-fluorouracil [5-FU]) has not been widely adopted in North America and is likely due to the technical difficulties and inconvenience associated with infusional chemotherapy. This study will substitute the oral chemotherapy drug capecitabine for infusional 5-FU in addition to substituting intravenous cisplatin with carboplatin (ECC - epirubicin, carboplatin and capecitabine). It is hoped that these substitutions will not only reduce the typical ECF related adverse effects but also allow for a more convenient administration of outpatient chemotherapy. It is also hoped that the genetic correlates of this study may also identify specific populations that preferentially benefit from ECC treatment.

DETAILED DESCRIPTION:
Background Information:

Capecitabine is an orally administered systemic prodrug of 5'-deoxy-5-fluorouridine which is converted to 5-fluorouracil. Capecitabine is readily absorbed from the gastrointestinal tract and then hydrolyzed in the liver. Capecitabine has been studied in the treatment of gastric/gastroesophageal cancer in addition to a wide variety of other malignancies (e.g. GI, breast).

Objectives

Phase I:

Primary Objective:

* To define the maximum tolerated dose (MTD) of capecitabine with combined fixed doses of epirubicin and carboplatin in patients with advanced solid cancers. With the identification of the MTD, determination of the recommended phase II dose will be made and used to further evaluate the specific anti-tumor activity of ECC in unresectable locally advanced and/or metastatic gastric/gastroesophageal cancer.

Secondary Objectives:

* To describe the safety, toxicity profile, principle and dose-limiting toxicities (DLT) of ECC when given on this schedule; and
* To determine the pharmacokinetic behavior of capecitabine when given in combination with epirubicin and carboplatin as part of the ECC regimen.

Phase II:

Primary Objective

* To determine the anti-tumor activity of ECC when given at the RPTD in patients who have unresectable locally advanced and/or metastatic gastric/gastroesophageal cancer who have not received prior palliative chemotherapy.

Secondary Objectives

* To further characterize the toxicity profile of the ECC regimen;
* To determine time to progression, duration of response, and overall survival of patients on this study;
* To determine the effects of thymidylate synthase (TS) polymorphisms on both toxicities and efficacy of ECC in prospectively genotyped patients;
* To prospectively evaluate other potential pharmacogenetic correlates which may also play a role in augmenting toxicity, including MTHFR; and
* To assess effects of uridine glucuronosyltransferase 2B7 (UGT 2B7) polymorphisms on epirubicin metabolism.

Study Design:

This is a Phase I/II trial that will study the safety as well as the efficacy of the ECC combination chemotherapy regimen.

Epirubicin: will be administered as an IV push at a fixed dose of 50mg/m2 on day 1 - repeated every 21 days

Carboplatin: will be administered IV, at a fixed dose with an AUC of 5 (over a 1-hour infusion in 500ml of 5% dextrose) on day 1 - repeated every 21 days

Capecitabine: will be administered as a twice daily oral medication (variable dose for phase I portion of the trial, but fixed dose for phase II portion of the trial) for 14 consecutive days (days 1-14) - repeated every 21 days

For the phase I portion of the study cohorts of 3 patients will be treated at each of 3 pre-determined dose levels of capecitabine and monitored for toxicity:

* Dose level 1: 750 mg/m2 bid
* Dose level 2: 850 mg/m2 bid
* Dose level 3: 1000 mg/m2 bid
* Dose level 4+: 25% dose escalation (rounded to the nearest twice a day dosing).

Statistical Analysis

Phase I:

Summary statistics such as frequency and intensity of toxicity occurring at each dose level will be provided. The percentage of patients developing DLT at each dose level will be computed. The dose-toxicity curve can be estimated accordingly using either parametric or non-parametric methods.

Phase II: A Simon's optimal two-stage phase II study will be conducted in patients with unresectable locally advanced or metastatic gastric or gastro-esophageal cancer at the RPTD of the ECC regimen. A total sample size of 43 patients will be required, 13 in the first stage and 30 in the second stage, if criteria for second stage accrual are met. If <=3/13 patients respond, this is deemed to correspond with the initial rejection limit and no further patients will be enrolled. If >=4/13 patients respond, an additional 30 patients will be enrolled in the second stage (total sample size = 43). Further statistical details are specifically outlined in Section 8 of the protocol. The response rate, standard error and its 95% confidence intervals (CI) will be calculated under the binomial distribution model. The efficacy of the regimen will then be evaluated by comparing the point estimates and 95% CI with historical data. Potential covariates for response will also be identified and evaluated via the logistic regression model. Kaplan-Meier estimates will be computed to estimate the secondary endpoints such as time to progression and survival. Cox-regression model can be applied incorporating covariates in the model. Fisher's exact test will be applied to compare the response rates between the different genetic TS polymorphisms groupings.

Stopping Rules:

Treatment will be discontinued and the patient will come off the trial therapy due to severe intercurrent illness, disease progression, unacceptable toxicity, patient request to stop, and/or if the physician deems it in the best interest of patient to discontinue.

Inclusion/Exclusion Criteria

Patient Population:

Phase I - Histologically or cytologically confirmed solid tumor refractory to conventional cytotoxic anticancer therapy, or for which there are no standard therapies with a reasonable therapeutic index.

Phase II - Inoperable/unresectable locally advanced and/or metastatic, histologically (or cytologically) confirmed adenocarcinoma or undifferentiated carcinoma of the stomach or gastro-esophageal junction presenting for first line palliative systemic treatment. Prior adjuvant chemoradiotherapy for gastric or gastroesophageal junction adenocarcinoma is allowed as long as the patient has completed adjuvant therapy >= 6 months prior to study entry. Patients need to have at least one site of measurable disease as defined by RECIST criteria.

Inclusion:

In general, to participate in the study, patients must be 18 years or older, have an expected life expectancy of > 12 weeks, WHO performance status 0-2, LVEF by MUGA > 50%, adequate organ function: hematological (ANC > 1.5X 10^9/L, platelets > 100 x 10^9/L, hepatic (bilirubin < 1.5 x ULN, AST/ALT < 3 x ULN), renal (calculated creatinine clearance > 60 ml/min). Negative pregnancy test for females with child-bearing potential. Prior radiotherapy allowed but must be delivered to < 25% of bone marrow, must be completed > 4 weeks before study entry and patients must have recovered from all side effects of the radiotherapy. Radiation must not be delivered to the sole response indicator lesion, unless there is documented evidence of disease progression in that site after completion of radiation. Patients must be able to reliably tolerate and comply with oral/feeding tube administered medications (patients are considered eligible if the investigator deems that there is no malabsorption syndrome and no GI obstruction that would impair the delivery of orally administered chemotherapy). If patient has had prior anthracycline, cumulative dose must be < 300mg/m2 of doxorubicin or its equivalent.

Exclusion:

Patients currently enrolled in another clinical trial involving active cancer treatment. Treatment with doxorubicin > 300mg/m2 or its equivalent. Serious medical conditions including myocardial infarction within 6 months prior to entry, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, congestive heart failure, uncontrolled hypertension, uncontrolled psychotic disorders, serious active infections, uncontrolled diabetes or any other medical condition that might be aggravated by study treatment. Pre-existing neuropathy > grade 1, history of seizures or patients receiving anti-epileptic prophylaxis, active and or progressive brain or leptomeningeal metastasis, pregnant or lactating women, patients with evidence or recent history of drug or alcohol abuse, prior treatment with capecitabine or infusional 5-FU, known hypersensitivity to carboplatin, 5-FU, anthracyclines or known DPD deficiency. Patients that lack physical integrity of the GI tract leading to intestinal obstruction. Patients taking warfarin, Coumadin or other coumarin derivatives. Presence of any mentally incapacitating psychological condition.

Recruitment:

The expected total number of patients to be enrolled (phase I and II) is 65.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cancer
* Gastric or esophageal cancer
* Adequate organ function and bone marrow reserve
* In general, patients must be 18 years or older
* Life expectancy of > 12 weeks
* World Health Organization (WHO) performance status 0-2
* Left ventricular ejection fraction (LVEF) by multiple gated acquisition (MUGA) > 50%
* Adequate organ function: hematological (ANC > 1.5 x 10^9/L; platelets > 100 x 10^9/L); hepatic (bilirubin < 1.5 x upper limit of normal [ULN]; AST/ALT < 3 x ULN); renal (calculated creatinine clearance > 60 ml/min).
* Negative pregnancy test for females with child-bearing potential
* Prior radiotherapy allowed but must be delivered to < 25% of bone marrow; must be completed > 4 weeks before study entry; and patients must have recovered from all side effects of the radiotherapy. Radiation must not be delivered to the sole response indicator lesion, unless there is documented evidence of disease progression in that site after completion of radiation.
* Patients must be able to reliably tolerate and comply with oral/feeding tube administered medications (patients are considered eligible if the investigator deems that there is no malabsorption syndrome and no gastrointestinal [GI] obstruction that would impair the delivery of orally administered chemotherapy).
* If patient has had prior anthracycline, cumulative dose must be < 300mg/m2 of doxorubicin or its equivalent.

Exclusion Criteria:

* Abnormal organ function or active infection
* Patients currently enrolled in another clinical trial involving active cancer treatment.
* Treatment with doxorubicin > 300mg/m2 or its equivalent.
* Serious medical conditions including myocardial infarction within 6 months prior to entry; unstable angina; active cardiomyopathy; unstable ventricular arrhythmia; congestive heart failure; uncontrolled hypertension; uncontrolled psychotic disorders; serious active infections; uncontrolled diabetes or any other medical condition that might be aggravated by study treatment.
* Pre-existing neuropathy > grade 1
* History of seizures or patients receiving anti-epileptic prophylaxis
* Active and or progressive brain or leptomeningeal metastasis
* Pregnant or lactating women
* Patients with evidence or recent history of drug or alcohol abuse
* Prior treatment with capecitabine or infusional 5-FU
* Known hypersensitivity to carboplatin
* 5-FU, anthracyclines or known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Patients that lack physical integrity of the gastrointestinal (GI) tract leading to intestinal obstruction.
* Patients taking warfarin (Coumadin) or other coumarin derivatives.
* Presence of any mentally incapacitating psychological condition.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-10; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
recommended phase II dose

SECONDARY OUTCOMES:
preliminary study of efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sawyer, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada